CLINICAL TRIAL: NCT04674332
Title: Comparative Study Between Use of Long Acting Insulin Versus Multiple Dose Regimen in Control of Gestational Diabetes Mellitus
Brief Title: Long Acting Insulin Versus Multiple Dose Regimen for Control of Gestational Diabetes Mellitus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maii medhat nawara, associate professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 323/2019
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Long Acting Insulin in Control of Gestational Diabetes Mellitus
MeSH Terms: interventions — Insulin, Long-Acting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- long acting insulin (Experimental)
  Interventions: Drug: Long acting insulin
- multiple dose regimen (Active Comparator)
  Interventions: Drug: multiple dose regimen

INTERVENTIONS:
Drug: Long acting insulin — long acting insulin analogue once daily at bed time
  Arms: long acting insulin
Drug: multiple dose regimen — intermediate and short acting insulin
  Arms: multiple dose regimen

SUMMARY:
multiple dose regimen as a standard treatment for gestational diabetes will be compared to long acting insulin

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with gestational diabetes mellitus
* between 24-28 weeks gestation

Exclusion Criteria:

* other endocrinological abnormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — they should be pregnant females
Enrollment: 148 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
time needed to achieve glycemic control | 1 year
  glycemic control assessed by fasting and postprandial blood sugar

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt